CLINICAL TRIAL: NCT03036813
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled, Multicenter Study of Voxelotor Administered Orally to Patients With Sickle Cell Disease
Brief Title: Study to Evaluate the Effect of Voxelotor Administered Orally to Patients With Sickle Cell Disease (GBT_HOPE)
Acronym: GBT_HOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GBT440-031; C5341043 (Other: Alias Study Number)
Expanded Access: NCT03943615 (No longer available)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Active Comparator): voxelotor
  Interventions: Drug: voxelotor
- Dose 2 (Active Comparator): voxelotor
  Interventions: Drug: voxelotor
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: voxelotor
  Other Names: GBT440
  Arms: Dose 1; Dose 2
Other: Placebo
  Arms: Placebo

SUMMARY:
A Phase 3, Double-blind, Randomized, Placebo-controlled, Multicenter Study of Voxelotor Administered Orally to Patients With Sickle Cell Disease

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double blind, parallel group, multicenter study of participants, age 12 to 65 years, with SCD. The key purpose for the study is to establish efficacy and safety of voxelotor as compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female study participants with sickle cell disease
2. Participants have had at least 1 episode of vaso-occlusive crisis (VOC) in the past 12 months.
3. Age 12 to 65 years
4. Hemoglobin (Hb) ≥5.5 and ≤10.5 g/dL during screening
5. For participants taking hydroxyurea (HU), the dose of HU (mg/kg) must be stable for at least 3 months prior to signing the ICF.

Exclusion Criteria:

1. More than 10 VOCs within the past 12 months that required a hospital, emergency room or clinic visit
2. Patients who are receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion) or have received a RBC transfusion for any reason within 60 days of signing the ICF
3. Hospitalized for sickle cell crisis or other vaso-occlusive event within 14 days of signing the ICF (i.e., a vaso-occlusive event cannot be within 14 days prior to signing the ICF)
4. Hepatic dysfunction characterized by alanine aminotransferase (ALT) >4 × upper limit of normal
5. Severe renal dysfunction (estimated glomerular filtration rate at the Screening visit; calculated by the central laboratory) <30 mL/min/1.73 m^2 or on chronic dialysis

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (28):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Little Rock, Arkansas
  - Oakland, California
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Newark, New Jersey
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Richmond, Virginia
- Toronto, Canada
- Egypt (3):
  - Alexandria
  - Cairo
  - Zagazig
- France (2):
  - Créteil
  - Paris
- Italy (3):
  - Monza, Milano
  - Padua
  - Verona
- Kingston, Jamaica
- Kenya (2):
  - Nairobi
  - Siaya
- Lebanon (2):
  - Beirut
  - Tripoli
- Netherlands (3):
  - Amsterdam
  - Rotterdam
  - The Hague
- Muscat, Oman
- Turkey (Türkiye) (3):
  - Adana
  - Kayseri
  - Mersin
- United Kingdom (2):
  - London
  - Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howard J, Ataga KI, Brown RC, Achebe M, Nduba V, El-Beshlawy A, Hassab H, Agodoa I, Tonda M, Gray S, Lehrer-Graiwer J, Vichinsky E. Voxelotor in adolescents and adults with sickle cell disease (HOPE): long-term follow-up results of an international, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Haematol. 2021 May;8(5):e323-e333. doi: 10.1016/S2352-3026(21)00059-4. Epub 2021 Apr 7. PMID 33838113
- [Derived] Minniti CP, Knight-Madden J, Tonda M, Gray S, Lehrer-Graiwer J, Biemond BJ. The impact of voxelotor treatment on leg ulcers in patients with sickle cell disease. Am J Hematol. 2021 Apr 1;96(4):E126-E128. doi: 10.1002/ajh.26101. Epub 2021 Feb 19. No abstract available. PMID 33476432
- [Derived] Vichinsky E, Hoppe CC, Ataga KI, Ware RE, Nduba V, El-Beshlawy A, Hassab H, Achebe MM, Alkindi S, Brown RC, Diuguid DL, Telfer P, Tsitsikas DA, Elghandour A, Gordeuk VR, Kanter J, Abboud MR, Lehrer-Graiwer J, Tonda M, Intondi A, Tong B, Howard J; HOPE Trial Investigators. A Phase 3 Randomized Trial of Voxelotor in Sickle Cell Disease. N Engl J Med. 2019 Aug 8;381(6):509-519. doi: 10.1056/NEJMoa1903212. Epub 2019 Jun 14. PMID 31199090
- [Derived] Metcalf B, Chuang C, Dufu K, Patel MP, Silva-Garcia A, Johnson C, Lu Q, Partridge JR, Patskovska L, Patskovsky Y, Almo SC, Jacobson MP, Hua L, Xu Q, Gwaltney SL 2nd, Yee C, Harris J, Morgan BP, James J, Xu D, Hutchaleelaha A, Paulvannan K, Oksenberg D, Li Z. Discovery of GBT440, an Orally Bioavailable R-State Stabilizer of Sickle Cell Hemoglobin. ACS Med Chem Lett. 2017 Jan 23;8(3):321-326. doi: 10.1021/acsmedchemlett.6b00491. eCollection 2017 Mar 9. PMID 28337324
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 449 subjects were screened for this study at 60 study sites. Between January 2017 and May 2018, a total of 274 subjects were randomized at 58 study sites across 12 countries. All 274 randomized subjects were included in the ITT Population. A total of 271 subjects received study drug and were included in the Safety Population.
Pre-assignment Details: Screening procedures were done within 35 days of randomization to assess eligibility.
Groups:
- Voxelotor 900mg: Participants received voxelotor 900 mg; administered orally, once daily for 72 weeks.
- Voxelotor 1500mg: Participants received voxelotor 1500 mg administered orally, once daily for 72 weeks.
- Placebo: Matching placebo; administered orally, once daily for 72 weeks.
Period: Overall Study
Arm/Group | Voxelotor 900mg | Voxelotor 1500mg | Placebo
Started | 92 | 90 | 92
Completed | 70 | 63 | 66
Not Completed | 22 | 27 | 26
Not completed — Adverse Event | 6 | 11 | 6
Not completed — Withdrawal by Subject | 12 | 6 | 10
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 1
Not completed — Non-Compliance | 1 | 5 | 3
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Other | 0 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Voxelotor 1500mg: Participants received voxelotor 1500 mg; administered orally, once daily for 72 weeks
- Total: Total of all reporting groups
Arm/Group | Voxelotor 900mg | Voxelotor 1500mg | Placebo | Total
Number analyzed (Participants) | 92 | 90 | 92 | 274
Age, Customized [Count of Participants; unit: Participants]
  12 to < 18 | 15 | 14 | 17 | 46
  >=18 to < 65 | 77 | 76 | 75 | 228
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 58 | 50 | 159
  Male | 41 | 32 | 42 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 10
  Not Hispanic or Latino | 86 | 82 | 85 | 253
  Unknown or Not Reported | 2 | 5 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Arab/Middle Eastern | 19 | 15 | 18 | 52
  Race: Black or African American | 60 | 59 | 63 | 182
  Race: White | 6 | 7 | 3 | 16
  Race: Asian | 0 | 1 | 0 | 1
  Race: Other | 4 | 2 | 5 | 11
  Race: Multiple | 2 | 5 | 3 | 10
  Race: Missing/ Not Specified | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Europe | 19 | 19 | 18 | 56
  North America | 36 | 34 | 35 | 105
  Egypt | 15 | 16 | 13 | 44
  Kenya | 17 | 14 | 18 | 49
  Jamaica | 0 | 2 | 2 | 4
  Oman | 2 | 2 | 5 | 9
  Lebanon | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Increase in Hb >1 g/dL From Baseline to Week 24
Description: Number of participants with increase in Hb >1 g/dL from Baseline to Week 24
Time Frame: Baseline to Week 24
Population: All randomized subject (ITT population).
Measure: Count of Participants; unit: Participants
Groups:
- Voxelotor 900 mg: Participants received voxelotor 900 mg administered orally, once daily
- Voxelotor 1500 mg: Participants received voxelotor 1500mg; administered orally, once daily
- Placebo: Participants received matching placebo; administered orally, once daily
Arm/Group | Voxelotor 900 mg | Voxelotor 1500 mg | Placebo
Number analyzed (Participants) | 92 | 90 | 92
Participants | 30 | 46 | 6

2. Secondary Outcome: Annualized Vaso-Occlusive Crisis (VOC) Incidence Rate
Description: Number of Vaso-Occlusive Crisis (VOC) events averaged per year.
Time Frame: Baseline to Week 72
Population: Population excludes 3 subjects (1 in the placebo group and 2 in the voxelotor 1500-mg group) who were not treated.
Measure: Mean (95% Confidence Interval); unit: Events per year
Groups:
- Voxelotor 900 mg: Participants received voxelotor 900 mg; administered orally, once daily
- Voxelotor 1500 mg: Participants received voxelotor 1500 mg; administered orally, once daily
Arm/Group | Voxelotor 900 mg | Voxelotor 1500 mg | Placebo
Number analyzed (Participants) | 92 | 88 | 91
Events per year | 2.4 [1.9 to 3.1] | 2.4 [1.8 to 3.1] | 2.8 [2.2 to 3.6]

3. Secondary Outcome: Percentage Change From Baseline in Hemolysis Measures
Description: Percentage change from Baseline to week 24 in unconjugated bilirubin
Time Frame: Baseline to Week 24
Population: Analysis population includes all randomized patients with a baseline value and at least one post-baseline value
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Voxelotor 900 mg | Voxelotor 1500 mg | Placebo
Number analyzed (Participants) | 88 | 85 | 85
percentage change | -20.1 (3.41) | -29.1 (3.46) | -2.8 (3.51)

4. Secondary Outcome: Percentage Change From Baseline in Hemolysis Measures
Description: Percentage change from Baseline to week 24 in the absolute reticulocyte which is used to estimate the degree of effective erythropoiesis. This values is important in Sickle Cell Disease and was reported by the central laboratory.
Time Frame: Baseline to Week 24
Measure: Least Squares Mean (Standard Error); unit: percentage change
Groups:
- Placebo: Participants will receive matching placebo; administered orally, once daily
Arm/Group | Voxelotor 900 mg | Voxelotor 1500 mg | Placebo
Number analyzed (Participants) | 92 | 88 | 91
percentage change | 4.7 (5.13) | -6.4 (5.17) | 4.7 (5.19)

5. Secondary Outcome: Percentage Change From Baseline in Hemolysis Measures
Description: Percentage change from Baseline to week 24 in reticulocytes % which is a % of total Red Blood Cells (RBCs).
Time Frame: Baseline to Week 24
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | Voxelotor 900 mg | Voxelotor 1500 mg | Placebo
Number analyzed (Participants) | 92 | 88 | 91
Percentage Change | -1.4 (4.65) | -18.0 (4.70) | 6.8 (4.73)

6. Secondary Outcome: Percentage Change From Baseline in Hemolysis Measures
Description: Percentage change from Baseline to week 24 in Lactate Dehydrogenase (LDH)
Time Frame: Baseline to Week 24
Population: Analysis population includes all randomized patients with a baseline value and at least one post-baseline value
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | Voxelotor 900 mg | Voxelotor 1500 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 87
Percentage Change | 1.6 (3.68) | -4.6 (3.69) | 3.0 (3.75)

ADVERSE EVENTS:
Time Frame: 72 Weeks
Description: Non-sickle cell disease (Non-SCD) related Adverse Events.
Groups:
- Voxelotor 900 mg: Participants received voxelotor 900 mg, administered orally, once daily
- Voxelotor 1500 mg: Participants received voxelotor 1500 mg administered orally, once daily
Arm/Group | Voxelotor 900 mg | Voxelotor 1500 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/92 | 2/88 | 2/91
Serious Adverse Events (participants affected / at risk) | 20/92 | 25/88 | 23/91
Other Adverse Events (participants affected / at risk) | 85/92 | 85/88 | 81/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voxelotor 900 mg (N=92) | Voxelotor 1500 mg (N=88) | Placebo (N=91)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 3 (4) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Malaria (Infections and infestations) | 3 (5) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Reticulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure high output (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripherial swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic sequestration (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extemity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voxelotor 900 mg (N=92) | Voxelotor 1500 mg (N=88) | Placebo (N=91)
Headache (Nervous system disorders) | 20 (22) | 27 (33) | 23 (34)
Diarrhoea (Gastrointestinal disorders) | 17 (24) | 20 (22) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (24) | 18 (33) | 13 (17)
Nausea (Gastrointestinal disorders) | 17 (21) | 16 (21) | 9 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (25) | 15 (17) | 12 (16)
Anaemia (Blood and lymphatic system disorders) | 6 (9) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (15) | 13 (17) | 10 (12)
Vomiting (Gastrointestinal disorders) | 13 (20) | 11 (17) | 15 (24)
Abdominal pain upper (Gastrointestinal disorders) | 14 (19) | 8 (9) | 6 (10)
Constipation (Gastrointestinal disorders) | 9 (9) | 6 (7) | 9 (9)
Gastritis (Gastrointestinal disorders) | 5 (7) | 3 (8) | 4 (4)
Pain (General disorders) | 15 (27) | 15 (27) | 18 (22)
Fatigue (General disorders) | 13 (16) | 12 (14) | 12 (15)
Pyrexia (General disorders) | 10 (13) | 11 (13) | 4 (5)
Non-cardiac chest pain (General disorders) | 13 (15) | 9 (10) | 10 (10)
Ocular icterus (Hepatobiliary disorders) | 9 (15) | 6 (7) | 8 (14)
Upper respiratory tract infection (Infections and infestations) | 22 (26) | 12 (13) | 13 (18)
Urinary tract infection (Infections and infestations) | 5 (8) | 9 (10) | 13 (15)
Tonsillitis (Infections and infestations) | 3 (5) | 5 (7) | 8 (10)
Malaria (Infections and infestations) | 2 (5) | 5 (8) | 3 (6)
Influenza (Infections and infestations) | 4 (5) | 3 (3) | 5 (6)
Gastroenteritis (Infections and infestations) | 6 (6) | 2 (2) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (33) | 12 (19) | 19 (22)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (5) | 5 (9) | 8 (22)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 5 (5)
Dizziness (Nervous system disorders) | 8 (10) | 4 (4) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (10) | 10 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (9) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (9) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8) | 4 (4) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT03036813/Prot_001.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT03036813/SAP_000.pdf